CLINICAL TRIAL: NCT00004552
Title: Etiology and Treatment of Alcohol Dependence
Brief Title: Acamprosate Treatment: Mechanisms of Action
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: NIAAAOMA03510; P50AA003510 (NIH)
Record Dates: First submitted 2000-02-03; First posted 2000-02-04 (Estimated); Last update posted 2015-07-02 (Estimated); Status verified 2015-06

CONDITIONS: Alcoholism
MeSH Terms: conditions — Alcoholism | interventions — Acamprosate

INTERVENTIONS:
Drug: acamprosate (Campral)

SUMMARY:
This study will examine whether pretreatment with two doses of acamprosate for seven days prior to abstinence lessens the intensity of acute withdrawal from alcohol compared with a placebo. Subjects will be randomly assigned to receive either one of two doses of acamprosate or placebo for seven days. This will be followed by a four- day inpatient period when withdrawal will be monitored. Additional drinking information will be obtained at a three month followup interview.

ELIGIBILITY:
Inclusion Criteria:

* Meets criteria for alcohol abuse or dependence.
* Able to read English at 6th grade level or higher and to complete study evaluations.
* Average weekly alcohol consumption of standard drinks of at least 25 drinks for men and 20 drinks for women.
* No more than 3 days abstinence/week.

Exclusion Criteria:

* Current abuse or dependence on other substances, other than nicotine and marijuana.
* Positive test results for opiates, cocaine, benzodiazepines and barbiturates.
* Regular use of psychoactive drugs including anxiolytics and antidepressants.
* Psychiatrically disabled.
* Hepatocellular disease or a history of cirrhosis.
* Medical conditions that would prevent the consumption of alcohol, increase the risk of complicated alcohol withdrawal, or prevent the use of acamprosate such as a history of neurological trauma or disease, seizures, delirium, or hallucinations, hepatic, cardiovascular, metabolic, endocrine, gastrointestinal, or kidney disease.
* Individuals who have had any significant physical illnesses during the two weeks prior to receiving study medication or during the medication treatment period prior to the withdrawal study.
* Medically detoxified from alcohol more than once within the past five years.
* Alcohol withdrawal symptoms requiring management with benzodiazepines.
* Females who are pregnant, nursing or not using a reliable method of birth control.
* Individuals who are seeking alcohol treatment or have been in alcohol treatment within the past six months.
* Individuals who report disliking spirits and have taken investigational drug or naltrexone within 4 weeks immediately preceding admission to study.
* Individuals who report any daily drug use during the thirty days prior to randomization for the following: anxiolytics, beta blockers, central nervous system stimulants, hypnotics, non-therapeutic doses of neuroleptics and antidepressants, drugs with psychotropic activity or drugs which cause excessive sedation.
* Subjects who have donated blood within the past six weeks.

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120
Dates: Study Completion 2002-12

CONTACTS AND LOCATIONS:
Locations (1):
- Substance Abuse Treatment Unit, University of Connecticut, New Haven, Connecticut, United States